CLINICAL TRIAL: NCT05872074
Title: Immediate and Short Term Outcomes for Using Drug Coated Balloons in Treating Coronary Bifurcation Lesions
Acronym: DCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, ahmed hassan, Assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CardioAinShams
Record Dates: First submitted 2023-04-14; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Ischemia; Heart; Stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Angiography

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional balloon (No Intervention): patients Who will undergo conventional provisional stenting using standard technique with plain balloon angioplasty wire both branches, MV and SB, with two coronary guide wires. Main branch pre-dilation Side branch pre-dilation using ordinary balloon for the side branch) Main vessel stenting Proximal optimization technique (POT) of the main vessel stent
- Drug coated balloon (Experimental): patients Who will undergo provisional stenting using Drug coated balloon (paclitaxel-coated balloon (PCB)) wire both branches, main vessel and side branch, with two coronary guide wires.
  Main branch pre-dilation Side branch pre-dilation using Drug coated balloon (paclitaxel-coated balloon for the side branch Main vessel stenting Proximal optimization technique (POT) of the main vessel stent
  Interventions: Diagnostic Test: Coronary angiography plus percutenous coronary intervention

INTERVENTIONS:
Diagnostic Test: Coronary angiography plus percutenous coronary intervention — 1. wire both branches, MV and SB, with two coronary guide wires.
  2. Main branch pre-dilation
  3. Side branch pre-dilation using (ordinary balloon in group "A" and Drug coated balloon in group "B" for the side branch)
  4. Main vessel stenting
  5. Proximal optimization technique (POT) of the main vessel stent
  Arms: Drug coated balloon

SUMMARY:
● the investigators aims to study the impact of using drug coated balloon in coronary artery bifurcation lesions on the procedural success rate & short-term MACE.

DETAILED DESCRIPTION:
Study Design:

A prospective study. Patients who met the inclusion criteria will be enrolled in our study will be subdivided into 2 groups :-

Group A: patient Who will undergo conventional provisional stenting using standard technique with plain balloon angioplasty Group B: patient Who will undergo provisional stenting using Drug coated balloon The patients will be randomly assigned for each group using a computer randomizing software application.

Both group with pass 3 stages: - Pre-procedural Interventional procedure Post -procedural Pre- procedural

History taking:

Age & sex. Family history. Smoking status. Medical history including hypertension (HTN), diabetes mellitus (DM), renal impairment, etc.

Previous history of coronary artery disease, myocardial infarctions (MI), revascularization procedures Medical treatment and any significant history of allergy Previous intervention history regarding (site, type, diameter and length of the stent , complications and TIMI flow ) if available

General &Physical examination:

with special emphasis on vital data, decubitus ,lung osculation and peripheral pulsation

Laboratory investigations:

Including kidney function, complete blood count, and High sensitive troponin in case of acute coronary syndrome Echocardiography will be done routinely for all patients with special emphasis on ejection fraction (to be assessed by modified Simpson's method), left ventricular dimensions, resting segmental wall motion abnormalities (RSWMAs).

Interventional procedure. Angiographic analysis. Serial coronary angiography will be performed at baseline (before and after intervention) and angiograms will be obtained in multiple views after intra-coronary nitrate if coronary spasm is suspected. coronary angiograms will be digitally recorded and analyzed by experienced personnel using a validated offline quantitative angiographic system and the following data will be collected: -

Bifurcation lesion distribution:

Left main artery bifurcation Left anterior descending artery/diagonal bifurcation Left circumflex artery/obtuse marginal bifurcation Right coronary artery/posterolateral branch

Medina classification the investigators will use Medina classification for coronary bifurcation lesion in which recording any narrowing more than 50% in each of the three arterial segments of the bifurcation in the following order: proximal main vessel (PMV). Distal main branch (DMV). Side branch (SB)

(1) is used to indicate the presence of a significant stenosis and (0) the absence of stenosis

Main vessel

Proximal reference diameter (mm) Distal reference diameter (mm) Mean reference diameter (mm) Minimal lumen diameter (mm) Percentage diameter stenosis (%)) Lesion length (mm) Angiographic restenosis (%)

Side branch

Reference diameter (mm) Minimal lumen diameter (mm) Percentage diameter stenosis (%) Lesion length (mm)

Type of drug-eluting stents Sirolimus-eluting stents Everolimus-eluting stents Zotrolimus-eluting stents Biolimus A9-eluting stent Number of stent/drug-eluting balloon used Stent/drug-eluting balloon size (mm) Stent/drug-eluting balloon length (mm) Maximum balloon size (mm) Maximum inflation pressure (atmosphere) other coronary lesions

Intervention

1. wire both branches, MV and SB, with two coronary guide wires.
2. Main branch pre-dilation
3. Side branch pre-dilation using (ordinary balloon in group "A" and Drug coated balloon in group "B" for the side branch)
4. Main vessel stenting
5. Proximal optimization technique (POT) of the main vessel stent

The following data will be recorded: -

1. Inflation time (Seconds.)
2. Inflation pressure (atmospheric pressure.)
3. Diameter of the stent after inflation
4. Time of the procedure After Intervention

1) Reference luminal diameter (mm) 2) Minimal luminal diameter in stent (mm) 3) Minimal luminal diameter in lesion (mm) 4) lesion success (attainment of >50% residual stenosis of the target lesion, as measured by quantitative coronary angiographic analysis) 5) procedure success (attainment of a final lesion success and no major angiographic complications as dissection or perforation ).

Post-procedural Medications will be prescribed according to 2018 ESC myocardial revascularization guidelines.

Patients will be assessed for immediate outcomes:

lesion success attainment of >50% residual stenosis of the target lesion, as measured by quantitative coronary angiographic analysis procedure success attainment of a final lesion success and no major complication as :-

A. Perforation with or without tamponade B. vascular access complications C. myocardial infarction D. contrast-induced nephropathy E. urgent coronary artery bypass grafting F. urgent repeat PCI G. Death.

Patients be assessed and monitor for 24 hours after the procedure and in the outpatient clinic after 6 months.

Follow up clinically after 6 months for MACEs

Study end points. Primary end point target is 6-month follow-up for:-

MACEs (major adverse cardiac events) defined as :-

1. Death
2. Non-fatal myocardial infarction
3. Target lesion re-vascularization (TLR) "defined as any clinically driven intervention (surgical or percutaneous) to the target lesion or any segment of the epicardial coronary artery containing the target lesion"
4. Stroke

Improvement or recurrence of symptoms (chest pain and dyspnea) Symptomatic patients will undergo coronary angiography and those who has no symptoms with undergo functional assessment using either (High dose dobutamine echo or Myocardial perfusion imaging )

Secondary end points included:

lesion success procedure success

ELIGIBILITY:
Inclusion criteria:

1. Patients with age above 18 years indicated for elective coronary angiography according to ESC 2018 guidelines with a bifurcation lesion affected Side branch (SB)
2. Patient Who planned for provisional stenting technique from the start or shifted to 2-stent strategy as a bailout to the Side branch
3. Bifurcation lesion with medina classification (1,1,1), (1,0,1) and (0,1,1)

Exclusion criteria:

Angiographical exclusion criteria as follows

1. Medina classification (1,1,0) or (0,1,0) or (1,0,0)
2. Side branch less than 2 mm in diameter
3. Patients who have multiple lesions with high syntax score and clinical characteristics favoring coronary artery bypass grafting according to latest ESC guidelines 2018.
4. Need for concomitant valvular surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-04 (Estimated); Primary Completion 2023-10-11 (Estimated); Study Completion 2023-10-11 (Estimated)

PRIMARY OUTCOMES:
MACE (Number of participants complains of one of MACE ) | 6 monthes
  Primary end point target is 6-month follow-up for:-
  o MACEs (major adverse cardiac events) defined as :-
  1. Death. (Measured as death or No death)
  2. Non-fatal myocardial infarction (defined according to ESC guidelines as the presence of acute myocardial injury detected by abnormal cardiac biomarkers in the setting of evidence of acute myocardial ischemia ). Measured as occurrence of events or not
  3. Target lesion re-vascularization (TLR) "defined as any clinically driven intervention (surgical or percutaneous) to the target lesion or any segment of the epicardial coronary artery containing the target lesion". Measured as need of revascularization by percutenous coronary intervention or coronary artery bypass grafting or not
  4. Stroke (loss of blood flow to part of the brain, which damages brain tissue transiently or permanently approved by clinical symptoms and imaging ( confirmed by CT or MRI) measured by occurrence of stroke or not

SECONDARY OUTCOMES:
Lesion and procedure | 6 monthes
  lesion success (Measured by attainment of >50% in- stent residual stenosis of the target lesion, as measured by quantitative coronary angiographic analysis) Attainment >50 % = 0 For 10% to 50 % = 1 Less than 10% = 2
  - procedure success (Measured as attainment of a final lesion success > 50% and no major complications as dissection or perforation ) No complication = 0 Any major complication= 1 . Each participants will take (0), (1) or (2) for each outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassan, MSc, Principal Investigator — Ain shams university , cardiology department
Locations (1):
- Ainshams university , Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Behan MW, Holm NR, de Belder AJ, Cockburn J, Erglis A, Curzen NP, Niemela M, Oldroyd KG, Kervinen K, Kumsars I, Gunnes P, Stables RH, Maeng M, Ravkilde J, Jensen JS, Christiansen EH, Cooter N, Steigen TK, Vikman S, Thuesen L, Lassen JF, Hildick-Smith D. Coronary bifurcation lesions treated with simple or complex stenting: 5-year survival from patient-level pooled analysis of the Nordic Bifurcation Study and the British Bifurcation Coronary Study. Eur Heart J. 2016 Jun 21;37(24):1923-8. doi: 10.1093/eurheartj/ehw170. Epub 2016 May 8. PMID 27161619
- [Background] Bukka M, Rednam PJ, Sinha M. Drug-eluting balloon: design, technology and clinical aspects. Biomed Mater. 2018 Feb 23;13(3):032001. doi: 10.1088/1748-605X/aaa0aa. PMID 29227279
- [Background] Hildick-Smith D, de Belder AJ, Cooter N, Curzen NP, Clayton TC, Oldroyd KG, Bennett L, Holmberg S, Cotton JM, Glennon PE, Thomas MR, Maccarthy PA, Baumbach A, Mulvihill NT, Henderson RA, Redwood SR, Starkey IR, Stables RH. Randomized trial of simple versus complex drug-eluting stenting for bifurcation lesions: the British Bifurcation Coronary Study: old, new, and evolving strategies. Circulation. 2010 Mar 16;121(10):1235-43. doi: 10.1161/CIRCULATIONAHA.109.888297. Epub 2010 Mar 1. PMID 20194880
- [Background] Cortese B, Bertoletti A. Paclitaxel coated balloons for coronary artery interventions: a comprehensive review of preclinical and clinical data. Int J Cardiol. 2012 Nov 1;161(1):4-12. doi: 10.1016/j.ijcard.2011.08.855. Epub 2011 Sep 28. PMID 21955612
- [Background] Jeger RV, Eccleshall S, Wan Ahmad WA, Ge J, Poerner TC, Shin ES, Alfonso F, Latib A, Ong PJ, Rissanen TT, Saucedo J, Scheller B, Kleber FX; International DCB Consensus Group. Drug-Coated Balloons for Coronary Artery Disease: Third Report of the International DCB Consensus Group. JACC Cardiovasc Interv. 2020 Jun 22;13(12):1391-1402. doi: 10.1016/j.jcin.2020.02.043. Epub 2020 May 27. PMID 32473887
- [Background] Khan MA, Hashim MJ, Mustafa H, Baniyas MY, Al Suwaidi SKBM, AlKatheeri R, Alblooshi FMK, Almatrooshi MEAH, Alzaabi MEH, Al Darmaki RS, Lootah SNAH. Global Epidemiology of Ischemic Heart Disease: Results from the Global Burden of Disease Study. Cureus. 2020 Jul 23;12(7):e9349. doi: 10.7759/cureus.9349. PMID 32742886
- [Background] Wilensky RL, Selzer F, Johnston J, Laskey WK, Klugherz BD, Block P, Cohen H, Detre K, Williams DO. Relation of percutaneous coronary intervention of complex lesions to clinical outcomes (from the NHLBI Dynamic Registry). Am J Cardiol. 2002 Aug 1;90(3):216-21. doi: 10.1016/s0002-9149(02)02457-8. PMID 12127606
- [Background] Rittger H, Brachmann J, Sinha AM, Waliszewski M, Ohlow M, Brugger A, Thiele H, Birkemeyer R, Kurowski V, Breithardt OA, Schmidt M, Zimmermann S, Lonke S, von Cranach M, Nguyen TV, Daniel WG, Wohrle J. A randomized, multicenter, single-blinded trial comparing paclitaxel-coated balloon angioplasty with plain balloon angioplasty in drug-eluting stent restenosis: the PEPCAD-DES study. J Am Coll Cardiol. 2012 Apr 10;59(15):1377-82. doi: 10.1016/j.jacc.2012.01.015. Epub 2012 Feb 29. PMID 22386286
- [Background] Niemela M, Kervinen K, Erglis A, Holm NR, Maeng M, Christiansen EH, Kumsars I, Jegere S, Dombrovskis A, Gunnes P, Stavnes S, Steigen TK, Trovik T, Eskola M, Vikman S, Romppanen H, Makikallio T, Hansen KN, Thayssen P, Aberge L, Jensen LO, Hervold A, Airaksinen J, Pietila M, Frobert O, Kellerth T, Ravkilde J, Aaroe J, Jensen JS, Helqvist S, Sjogren I, James S, Miettinen H, Lassen JF, Thuesen L; Nordic-Baltic PCI Study Group. Randomized comparison of final kissing balloon dilatation versus no final kissing balloon dilatation in patients with coronary bifurcation lesions treated with main vessel stenting: the Nordic-Baltic Bifurcation Study III. Circulation. 2011 Jan 4;123(1):79-86. doi: 10.1161/CIRCULATIONAHA.110.966879. Epub 2010 Dec 20. PMID 21173348
- [Background] Niccoli G, Ferrante G, Porto I, Burzotta F, Leone AM, Mongiardo R, Mazzari MA, Trani C, Rebuzzi AG, Crea F. Coronary bifurcation lesions: to stent one branch or both? A meta-analysis of patients treated with drug eluting stents. Int J Cardiol. 2010 Feb 18;139(1):80-91. doi: 10.1016/j.ijcard.2008.10.016. Epub 2008 Nov 22. PMID 19027969
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO. 2018 ESC/EACTS Guidelines on myocardial revascularization. EuroIntervention. 2019 Feb 20;14(14):1435-1534. doi: 10.4244/EIJY19M01_01. No abstract available. PMID 30667361
- [Result] Ann SH, Balbir Singh G, Lim KH, Koo BK, Shin ES. Anatomical and Physiological Changes after Paclitaxel-Coated Balloon for Atherosclerotic De Novo Coronary Lesions: Serial IVUS-VH and FFR Study. PLoS One. 2016 Jan 29;11(1):e0147057. doi: 10.1371/journal.pone.0147057. eCollection 2016. PMID 26824602